CLINICAL TRIAL: NCT02814812
Title: Postoperative Comput Tomography as a Predictor of Postoperative Complications After Pancreatic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PO14086
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2019-12

CONDITIONS: Pancreatectomy

ARMS (1):
- pancreatic surgery (Experimental)
  Interventions: Procedure: CT scan

INTERVENTIONS:
Procedure: CT scan

SUMMARY:
Pancreatectomy represents the classic approach for resectable lesions of the pancreas, duodenum and periampullary region. Due to the technical skills required, the complex anatomy and the extreme fragility of the pancreatic parenchyma, pancreatic resection is still considered to be at risk of postoperative complication mainly due to pancreatic juice leaks. Anastomotic leaks are the major cause of morbidity and in-hospital mortality due to the activation of pancreatic enzymes and the following infectious and hemorrhagic complications. Severe complications negatively affect postoperative outcomes, long-term survival, quality of life, and costs. Operative mortality traditionally has been defined as the rate within 30 days or during the initial hospitalization. But in pancreatic surgery mortality rates within 90 days after pancreatic resection are double those at 30 days. In the present study, the investigators sought to evaluate the usefulness of postoperative CT-scan on the seventh postoperative day before discharging the patients to detect undiagnosed postoperative complication.

ELIGIBILITY:
Inclusion Criteria:

Will be included in this study, patients:

* Having an indication of pancreatic surgery
* In scheduled surgery
* Agreeing to participate in the research (ie who signed the informed consent to research participation)
* >18yo

Exclusion Criteria:

Will not be included in this study, patients:

* With emergency surgery
* Protected by law
* Under 18 years
* Presenting an against-indications to the scanner: documented severe allergy to contrast material, kidney failure against-showing the contrast medium injection, pregnancy, lactation and/or MRI (pacemaker, metallic intraocular foreign body)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
detection of undiagnosed postoperative complication by CT scan | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Background] Durot C, Rousset P, Thivolet A, Passot G, Deguelte S, Dohan A, Glehen O, Hoeffel C. What the radiologist should know about postoperative MDCT evaluation of a patient treated with cytoreductive surgery with or without hyperthermic intraperitoneal chemotherapy. Clin Radiol. 2018 Jun;73(6):517-525. doi: 10.1016/j.crad.2018.02.001. Epub 2018 Mar 21. PMID 29573786